CLINICAL TRIAL: NCT01926938
Title: Endothelial Function in Young Hispanic Adults at Risk for Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Enrique Caballero, Clinical Investigator/Director, Latino Diabetes Initiative, Joslin Diabetes Center
Other Study IDs: CHS#: 03-30
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- adults at risk: Latino adults with family history of type 2 diabetes
- controls: Latino adults without family history of type 2 diabetes and normal glucose tolerance

SUMMARY:
Diabetes is a major public health problem. Hispanics/Latinos are known to be at higher risk for type 2 diabetes. The function of the endothelium has played a key role in the understanding of vascular complications in people with diabetes. Endothelial function and vascular reactivity are impaired not only in white adults with type 2 diabetes but also in those at risk for the disease by virtue of having impaired glucose tolerance or parental history of type 2 diabetes. Whether this finding is applicable to hispanics is not known. The investigators plan to assess the endothelial function and vascular reactivity in young Hispanic adults at risk of developing type 2 diabetes by virtue of being obese and belonging to a minority population.

ELIGIBILITY:
Inclusion Criteria:

* Group 1:

  1. Age between 18-40 years;
  2. Hispanic (we will consider a subject being Hispanic if both parents are reported as Hispanics when asked the following question: "What ethnic group do you consider that you belong to?");
  3. History of type 2 diabetes in one or both parents;
  4. BMI above 27;
  5. Not have participated in any exercise program for the 6 months prior to the beginning of the study.

Group 2:

1. Age between 18-40 years;
2. Hispanic (same criteria as above );
3. No history of type 2 diabetes in any first degree relative;
4. BMI under 25;
5. Not have participated in any exercise program for the 6 months prior to the beginning of the study.

Exclusion Criteria:

* diabetes, glucose intolerance, pregnancy, smoking, cardiovascular disease, uncontrolled hypertension, renal disease, proteinuria, cancer, infectious diseases, severe GI diseases, lung disease, electrolyte abnormalities, anemia, endocrine disorders, severe dyslipidemia, peripheral vascular disease, medications: beta-blockers, any diuretic, calcium channel blockers, ACE inhibitors, angiotensin receptor blockers, niacin, glucocorticoids, any antineoplastic agent, antibiotics, psychoactive agents, bronchodilators or insulin.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young Latino adults with and without family history of type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2003-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
markers of endothelial activation, coagulation and inflammation | cross sectional evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Caballero, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States